CLINICAL TRIAL: NCT04362553
Title: Advanced Wireless, Wearable Sensors for Continuous Hemodynamic Monitoring
Status: Completed | Type: Observational
Sponsor: Northwestern University (Other)
Responsible Party: Principal Investigator, Shuai (Steve) Xu, Principal Investigator, Northwestern University
Other Study IDs: STU00210413
Record Dates: First submitted 2020-04-15; First posted 2020-04-27 (Actual); Last update posted 2022-09-28 (Actual); Status verified 2022-09

CONDITIONS: Congestive Heart Failure
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Adults: Adults scheduled to receive a TTE (Trans-esophogeal echocardiogram)
  Interventions: Device: wearable vital signs sensor

INTERVENTIONS:
Device: wearable vital signs sensor — vital signs monitoring during standard of care procedures; TTE, swan-ganz catheterization

SUMMARY:
Percent agreement of vital signs monitoring between the experimental sensor and standard of care monitoring

ELIGIBILITY:
Inclusion Criteria

1. Patient's aged 18-65
2. Patient's scheduled to undergo a Trans-thoracic Echocardiogram (TTE) in an outpatient cardiology clinic or admitted to the Cardiac Care Unit with a swan ganz catheter in place for continuous invasive hemodynamic monitoring

Exclusion Criteria

1. Patient's with fragile skin or skin conditions that would prevent them from having a sensor placed
2. Patients undergoing exercise or drug induced cardiac stress test
3. Patients with a visible wound at site of sensor placement 3.4. Patients with structural or functional limitations to peripheral blood flow (known upper extremity peripheral arterial disease, use of vasopressors etc.).

Ages: 18 Years to 65 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Cardiology patients
Sampling Method: Non-Probability Sample
Enrollment: 42 (Actual)
Dates: Start 2020-06-01 (Actual); Primary Completion 2020-11-23 (Actual); Study Completion 2022-09-05 (Actual)

PRIMARY OUTCOMES:
Percent agreement with pilot sensor and current standard of vital signs monitoring | 2 years
  Percent agreement with pilot sensor and current standard of vital signs monitoring

CONTACTS AND LOCATIONS:
Locations (1):
- Northwestern Memorial Hospital, Chicago, Illinois, United States

IPD SHARING:
Plan to Share IPD: No